CLINICAL TRIAL: NCT04120948
Title: Laser Tongue Debridement for Oral Malodor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Head & Neck Institute (Other)
Collaborators: Biolase Inc (Industry); Ohio State University (Other)
Responsible Party: Principal Investigator, victor kizhner, MD, New York Head & Neck Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NY Head and Neck
Record Dates: First submitted 2019-09-25; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Waterlase Express Laser System (Experimental): 10-minute treatment with the Waterlase Express (Biolase, Irvine CA). The dorso-posterior surface of the tongue is treated with the laser in 10 passes of 60 seconds each with 10 seconds of rest in between. Laser settings were 60μs pulse width, 4W, 40Hz, 10% air and 5% water irrigation. An MC12 sapphire laser tip (Biolase, Irvine CA) is held 3mm away from the tongue in a constant sweeping motion during treatment with passes overlapping passes in alternate direction, side to side motion and front to back motion with laser fluence on the tongue surface calculated at 3J/cm2. The settings were non ablative and non thermal.
  Interventions: Device: Waterlase Express Laser System
- Tongue scraper (Active Comparator): tongue scraping
  Interventions: Device: Tongue scraper

INTERVENTIONS:
Device: Waterlase Express Laser System — 10-minute treatment with the Waterlase Express (Biolase, Irvine CA). The dorso-posterior surface of the tongue is treated with the laser in 10 passes of 60 seconds each with 10 seconds of rest in between. Laser settings were 60μs pulse width, 4W, 40Hz, 10% air and 5% water irrigation. An MC12 sapphire laser tip (Biolase, Irvine CA) is held 3mm away from the tongue in a constant sweeping motion during treatment with passes overlapping passes in alternate direction, side to side motion and front to back motion with laser fluence on the tongue surface calculated at 3J/cm2. The settings were non ablative and non thermal.
  Arms: Waterlase Express Laser System
Device: Tongue scraper — mechanical scraping of the dorso-posterior surface of the tongue
  Arms: Tongue scraper

SUMMARY:
Malodor is a multifactorial condition with oral pathology representing the main culprit and the tongue being the first to second contributor to the malodor. Bacterial load can represent a quantifiable measure regardless of the original pathology. It is hypothesized that reduction in malodor can be represented by tongue changes both in appearance, bacterial and biofilm load reduction (measured by CFU and volatile gases measurement), organoleptic measurement and subjective improvement.

Methods: A randomized controlled prospective study under IRB approval. Diagnostic criteria for enrollment and follow up were organoleptic test by 2 judges, halimeter reading, tongue colores changes HALT questionnaire and direct aerobic and anaerobic tongue cultures measured by CFU. Patients were treated with laser tongue debridement (LTD) with an Er,Cr:YSGG solid state laser has been shown to be effective in biofilm reduction.

ELIGIBILITY:
Inclusion Criteria:

* an individual (male or female) who can understand and voluntarily sign an informed consent form
* a baseline organoleptic oral malodor score of at least 2

Exclusion Criteria:

* severe caries,
* signs of gingival inflammation on intraoral exam
* possible extra-oral halitosis (tonsillitis, sinusitis, and pulmonary pathologic conditions, or a condition that may contribute to systemic halitosis, such as hepatic cirrhosis or uncontrolled diabetes)
* antibiotic treatment within 1 month prior to study
* pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Halimeter measurement | change from baseline to 1 month
  Measurement of volatile sulfur compounds in patient's breath.

SECONDARY OUTCOMES:
HALT questionnaire | change from baseline to 1 month
  Quality of life (QOL) questionnaire that ranks responses. The total score is evaluated on a scale of 0-100. A score of 0 correlates to no perceived effect on QOL, and a score of 100 correlates to a severe perceived effect on QOL.

OTHER OUTCOMES:
bacterial load | change from baseline to 1 month
  Sample is collected from the dorsal tongue surface. Total anaerobic and aerobic bacterial colonies are counted (CFU).

CONTACTS AND LOCATIONS:
Locations (1):
- New York Head & Neck Institute offices, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krespi YP, Kizhner V, Wilson KA, Sivriver A, Low S, Khosravi Y, Stoodley P. Laser tongue debridement for oral malodor-A novel approach to halitosis. Am J Otolaryngol. 2021 Jan-Feb;42(1):102458. doi: 10.1016/j.amjoto.2020.102458. Epub 2020 Mar 13. PMID 33045536